CLINICAL TRIAL: NCT01240122
Title: Short-Term Evaluation of Corneal Staining With Balafilcon A Lenses and Two Multi-Purpose Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: COBR-109-9608
Record Dates: First submitted 2010-11-08; First posted 2010-11-15 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Corneal Staining
Keywords: Corneal staining and comfort evaluation in normal, habitual contact lens wearers.

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Biotrue MPS (Active Comparator)
  Interventions: Device: Biotrue MPS
- Investigational MPS (Experimental)
  Interventions: Device: Investigational MPS

INTERVENTIONS:
Device: Biotrue MPS — Multi-purpose contact lens care solution
  Arms: Biotrue MPS
Device: Investigational MPS — Multi-purpose contact lens care solution
  Arms: Investigational MPS

SUMMARY:
An investigational multi-purpose solution (MPS)was clinically evaluated against Biotrue MPS at specific time points over the course of four days. The study was conducted with PureVision lenses.

ELIGIBILITY:
Inclusion Criteria:

* were at least 18 years old;
* were experienced contact lens wearers;
* were correctable to at least 20/40 or better in both eyes with contact lenses;
* were in good general health, with healthy eyes (other than requiring vision correction);
* had not worn lenses for at least 12 hours before each baseline visit;
* had a corneal staining score no greater than Grade 1 in either eye at time of enrollment;
* had previously used an MPS or hydrogen peroxide solution successfully.

Exclusion Criteria:

* had a confirmed diagnosis of Sjögren's syndrome or other condition that results in a chronic and/or pathologic dry eye condition;
* required concurrent ocular medication or have used ocular medication within 24 hours of entering the study;
* had a known sensitivity or intolerance to any MPS, study products or ingredient(s);
* were currently participating in any other clinical study;
* had a condition or are in a situation that, in the investigator's opinion, may put them at significant risk, confound the study results, or interfere significantly with their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08-31 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Y Kao, OD, Principal Investigator — AMO
Locations (1):
- Abbott Medical Optics Inc, Santa Ana, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Biotrue/Investigational MPS: Paired/parallel eye evaluation; each subject used both study treatments and were tested at 1 hour, 2hours, 4 hours and end of day during a 4 day period.
Period: Overall Study
Arm/Group | Biotrue/Investigational MPS
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biotrue/Investigational MPS
Number analyzed (Participants) | 29
Age, Customized [Number; unit: participants]
  <18 years | 0
  18 years of age or older | 29
Sex/Gender, Customized [Number; unit: participants] — Gender was not an analysis endpoint for this study.
  participants
    Male | 0
    Female | 0
    Unknown | 29

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining by Wear Time
Description: All participants were contact lenses wearers and were evaluated with a Corneal Staining at 1 hour, 2 hours, 4 hours and end of day. The corneal staining test is performed using fluorescein drops in the eye and ultraviolet illumination to determine if there has been any damage to the cornea from the use of the lens solutions or from the use of the contact lens.
Time Frame: 1 hour on Day 1, 2 hours on Day 2, 4 hours on Day 3 and End of Day on Day 4
Population: Corneal Staining Severity at Scheduled Visits (Safety Population)
Measure: Number; unit: participants
Groups:
- Biotrue: Paired/parallel eye evaluation; each subject was treated with Biotrue, and were tested at 1 hour, 2 hours, 4 hours and end of day during a 4 day period.
- Investigational MPS: Paired/parallel eye evaluation; each subject used both used the Investigational MPS and were tested at 1 hour, 2 hours, 4 hours and end of day during a 4 day period.
Arm/Group | Biotrue | Investigational MPS
Number analyzed (Participants) | 29 | 29
participants
  Staining at 1 Hour, Day 1 | 19 | 15
  Staining at 2 Hours, Day 2 | 19 | 7
  Staining at 4 Hours, Day 3 | 21 | 5
  Staining at End of Day, Day 4 | 18 | 8

2. Secondary Outcome: Subjective Solution Preference
Description: All subjects were asked which solution they prefer based on comfort level: Biotrue MPS, Investigational MPS, or no difference.
Time Frame: Day 4
Population: All subjects who completed the study were included in the analysis per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Biotrue MPS: Paired/parallel eye evaluation; each subject was treated with Biotrue multi-purpose solution in one eye, and was tested at 1 hour, 2 hours, 4 hours and end of day during a 4 day period.
- Investigational MPS: Paired/parallel eye evaluation; each subject used Investigational MPS in the alternate eye and was tested at 1 hour, 2 hours, 4 hours and end of day during a 4 day period.
Arm/Group | Biotrue MPS | Investigational MPS
Number analyzed (Participants) | 28 | 28
Participants
  Subject preferred the solution | 6 | 7
  Subject did not prefer the solution | 7 | 6
  Subject reported solutions were about the same | 15 | 15

3. Secondary Outcome: Overall Ocular Comfort
Description: All subjects were asked to rate their lens comfort at each visit based on an 11 point scale where 0 meant that the lens could not be tolerated and 10 indicated that the lens could not be felt.
Time Frame: Day 4
Population: All subjects who completed the study were included in the analysis per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Biotrue: Paired/parallel eye evaluation; each subject was treated with Biotrue MPS in one eye, and was tested at 1 hour, 2 hours, 4 hours and end of day during a 4 day period.
- Investigational MPS: Paired/parallel eye evaluation; each subject used the Investigational MPS in the alternate eye, and was tested at 1 hour, 2 hours, 4 hours and end of day during a 4 day period.
Arm/Group | Biotrue | Investigational MPS
Number analyzed (Participants) | 29 | 29
score on a scale | 8.3 (1.74) | 8.4 (1.48)

ADVERSE EVENTS:
Arm/Group | Biotrue/Investigational MPS
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes